CLINICAL TRIAL: NCT06011421
Title: Wound Catheter Vs LA Bolus in Renal Transplant: RCT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: GS21/138922
Record Dates: First submitted 2023-08-21; First posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Wound
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Local Anaesthetic Wound Catheter Insertion — Use of the Local Anaesthetic Wound Catheter Insertion during kidney transplant

SUMMARY:
Pain control is an important part of patients' care after a kidney transplant. Currently patients receive a one off injection of Local Anaesthetic (LA) in the wound at the end of the operation followed by Intravenous morphine through a Patient Controlled Analgesia System (PCAS), a button pressed to provide a calculated dose with lock out times for safety.

Through this study the aim to test the efficiency of Continuous Local Anaesthetic Infiltration via Wound Catheter (LAWC) which is a method to deliver Local Anaesthetic over a longer period of time after the operation. LAWC are currently in use in a variety of surgical specialities including Liver surgery. Patients participating in this study will be allocated randomly to one of 2 groups; one will receive LA at the end of the operation as per current practice and one will receive LAWC. It then compare outcomes such as the the dose of morphine required in the PCAS, quality of pain control and improvement in recovery.

ELIGIBILITY:
Inclusion Criteria:

* Primary kidney transplantation
* Single kidney transplantation
* Signed informed Consent

Exclusion Criteria:

* Midline laparotomy
* Dual kidney transplantation
* Kidney re-transplantation
* Multi-organ transplantation
* Patients on Long term opiates
* Patients with psychiatric illness

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing kidney transplant
Sampling Method: Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2022-01-31 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Total Dose of IV Morphine in the first 24 hours post op | 24 hours
  Measurment of the dose delivered in 24 hours

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Leeds Teaching Hospital NHS Trust, Leeds
  - Leeds Teaching Hospitals NHS Trust, Leeds